CLINICAL TRIAL: NCT00688077
Title: Evaluation of FGF-23 Suppressibility by Calcitonin in Healthy Men - Pilot Study
Brief Title: FGF-23 Suppressibility by Calcitonin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: H. de Boer MD. PhD., Rijnstate Hospital, Arnhem
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LTC-524/030408
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Hypophosphatemia
Keywords: Fibroblast growth factor - 23; Calcitonin
MeSH Terms: conditions — Hypophosphatemia | interventions — Calcitonin

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Calcitonin
- 2 (Placebo Comparator): NaCl 0,9% 2 ml, single subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcitonin — Calcitonin 200 IU/ml, single subcutaneous injection, experimental group
  Arms: 1
Drug: Placebo — NaCl 0,9 % 1ml, single subcutaneous injection, placebo group
  Arms: 2

SUMMARY:
Introduction:

Based on our experience with calcitonin as an FGF-23 suppressive agent in a patient with an FGF-23 producing tumor we hypothesize that calcitonin may be a physiologically important regulator of FGF-23 production and secretion in healthy humans.

Aim:

In this study we wish to examine the FGF-23 suppressive effects of calcitonin in healthy men.

Study Design:

placebo-controlled, cross-over study

Method:

* All twelve subjects are examined on two occasions, once after exposure to placebo 1 ml NaCl 0.9% subcutaneously, and once following calcitonin 200 IU/ml subcutaneously
* On both occasions frequent bloodsampling will take place, out an indwelling catheter in de forearm vein.
* Sampling times: -15, 0, 60, 120, 240, 360, and 480 minutes
* Mealtimes: Calcium and Phosphate intake standardized on both occasions
* All samples are analyzed for FGF-23, using a C-terminal FGF-23 ELISA kit (Immunotopics, San Clemente, USA) that measures intact and C-terminal fragments of FGF-23, and one that measures only intact FGF-23
* Samples obtained at T-15, T0, T240 and T480 are stored for later analysis of Ca, albumin, PO4, PTH, 25-OHD and 1,25-OHD

Endpoint:

A change of 25% in de serum FGF-23 levels in response to a single subcutaneous injection of calcitonin 200 IU.

ELIGIBILITY:
Inclusion Criteria:

* Healthy man, who are between 20-55 years old, and have a BMI 20-27 kg/m2.

Exclusion Criteria:

* Serum creatinin >100 mmol/L, or glomerular filtration rate <80 ml/min.
* Abnormal serum Ca, PO4, albumin, 25-OH vitamin D, or PTH levels.
* Any medication.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2008-05; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
A change of 25% in de serum FGF-23 levels in response to a single subcutaneous injection of calcitonin 200 IU. | eight hours

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands